CLINICAL TRIAL: NCT01122212
Title: Introduction of Protein S100 in the Routine Diagnostics in Patients With Minor Head Injury
Brief Title: Introduction of Protein S100 in Diagnostics in Minor Brain Injury Patients at Our Hospital
Acronym: S100
Status: Completed | Type: Observational
Sponsor: Kantonsspital Münsterlingen (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: S100-01 2010
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2012-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; ct scans; protein s100; inpatient treatment
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood (Serum)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In Patients with minor head injury measurement of protein S100 will be introduced to the emergency departement as another tool to rule out intracerebral bleeding.

DETAILED DESCRIPTION:
Severe intracerebral bleeding is still a complication even in obvious minor head injury (MHI) that makes the use of CT scanning necessary in patients with only few signs of intracerebral injury. To reduce the number of cerebral CT scans without pathologic findings measurement of protein S100 level in serum will be used in the emergency departement (ED) at our hospital.

Our hypothesis: with measurement of S100 levels cCT scans and inpatient treatment can be reduced, radiation and costs can be reduced.

From January 1st 2010 for 3-6 months all patients with head injury (all GCS) will be tested for their initial S100 level. Cut off level is set at 0,105ng/ml. During this period test results will be blinded. Decisions for further diagnostics (x-ray, cCT) and inpatient vs. outpatient treatment are made on clinical impressions as they are made now. The test results will be monitored and compared with clinical cases. Sensitivity, specificity, positive and negative predictive values will be measured.

The aim is to identify patients without risk for intracerebral bleeding (ie S100 level lower than 0,105ng/ml). Those can be managed in an outpatient way. All other patients will be diagnosed and treated as it is now.

If the test will not miss one intracranial bleeding and will save cCT scans and inpatient treatment, measurement of protein S100 will become a routine diagnostic in our ED for patients with MHI.

ELIGIBILITY:
Inclusion Criteria:

* history of MHI during last 6 hours
* older than 3 years

Exclusion Criteria:

* more than 6 hours after MHI
* younger than 4 years
* informed consent not given

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients older than 3 years entering the ED of the Kantonsspital Münsterlingen with the history of a MHI during the last 6 hours and after getting informed consent
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Blay, MD, Principal Investigator — Kantonsspital Münsterlingen
Locations (1):
- Kantonsspital Münsterlingen, Münsterlingen, Thurgau, Switzerland